CLINICAL TRIAL: NCT05209295
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Pharmacokinetics of CC-486 (Onureg®) in Subjects With Moderate or Severe Hepatic Impairment Compared With Normal Hepatic Function in Adult Subjects With Myeloid Malignancies
Brief Title: A Study to Evaluate CC-486/Onureg in Participants With Moderate or Severe Hepatic Impairment Compared With Normal Hepatic Function in Participants With Myeloid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CA055-001
Expanded Access: NCT03723135 (Approved for marketing)
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Insufficiency; Neoplasms
Keywords: CC-486; Azacitidine; Hepatic Impairment; Onureg; Myeloid Malignancies
MeSH Terms: conditions — Hepatic Insufficiency; Neoplasms | interventions — cc-486; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental)
  Interventions: Drug: Onureg
- Group 2 (Experimental)
  Interventions: Drug: Onureg
- Group 3 (Other): Control - participants with normal hepatic function
  Interventions: Drug: Onureg

INTERVENTIONS:
Drug: Onureg — Specified dose on specified days
  Other Names: CC-486, Oral Azacitidine

SUMMARY:
The purpose of this study is to evaluate the effect of moderate or severe liver impairment on the drug levels of oral azacitidine and the safety and tolerability of oral azacitidine in participants with myeloid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Myelodysplastic syndrome, Acute myeloid leukemia, Non-acute promyelocytic leukemia, Chronic myelomonocytic leukemia, Philadelphia-negative myeloproliferative neoplasms, Myelodysplastic syndrome Myeloproliferative neoplasms overlap, Accelerated phase and blast phase Myeloproliferative neoplasms, Blastic plasmacytoid dendritic cell neoplasm according to the World Health Organization (WHO) 2016 classification
* Life expectancy of ≥ 3 months
* Stable renal function without dialysis for at least 2 months prior to investigational product administration
* Has moderate or severe hepatic impairment as defined by National Cancer Institute Organ Dysfunction Working Group criteria

Exclusion Criteria:

* Chemotherapy or radiotherapy within 2 weeks or 5 half-lives, whichever is longer, prior to the first day of investigational product administration
* Persistent, clinically significant non-hematologic toxicities from prior therapies which have not recovered to < Grade 2
* Any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study
* History of inflammatory bowel disease, celiac disease, prior gastrectomy, gastric bypass, upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption of the investigational product and/or predispose the participant to an increased risk of gastrointestinal toxicity

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
AUC0-t: Estimation of area under the plasma concentration-time curve (AUC) calculated from time zero to the last measured time point | Day 1
AUC0-∞: Estimation of AUC calculated from time zero to infinity | Day 1
Cmax: Observed maximum concentration | Day 1

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 9 Months
Incidence of serious adverse events | Up to 9 Months
Number of participants with clinically significant changes in electrocardiogram parameters | Up to 9 Months
Incidence of clinically significant changes in vital signs: Body temperature | Up to 9 Months
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 9 Months
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 9 Months
Incidence of clinically significant changes in vital signs: Heart rate | Up to 9 Months
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 9 Months
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 9 Months
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 9 Months
Number of Participants with clinically significant changes in Eastern Cooperative Oncology Group (ECOG) performance status | Up to 9 Months
Incidence of clinically significant changes in clinical laboratory results: Liver Function tests | Up to 9 Months
Number of clinically significant changes in physical examinations | Up to 9 Months
Number of participants with a recording of concomitant medications | Up to 9 Months
Number of participants with a recording of concomitant procedures | Up to 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- United States (4):
  - Local Institution - 0083, Iowa City, Iowa
  - Local Institution - 0069, Detroit, Michigan
  - Local Institution, Cleveland, Ohio
  - Local Institution - 9003, Charlottesville, Virginia
- Argentina (4):
  - Local Institution - 0011, Pilar, Buenos Aires
  - Local Institution - 0010, ABB, Buenos Aires F.D.
  - Local Institution - 0014, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0012, Buenos Aires
- Colombia (3):
  - Local Institution - 0085, Bogotá, Bogota D.C.
  - Local Institution - 0084, Bogota, Cundinamarca
  - Local Institution - 0086, Piedecuesta, Santander Department
- Germany (3):
  - Local Institution - 0076, Augsburg, Bavaria
  - Local Institution - 0075, Halle, Saxony-Anhalt
  - Local Institution - 0074, Hamburg
- Spain (4):
  - Local Institution - 0018, Badalona, Barcelona [Barcelona]
  - Local Institution - 0017, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0015, Pamplona, Navarre
  - Local Institution - 0078, Salamanca

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com